CLINICAL TRIAL: NCT03018613
Title: Evaluation of the Effect of Fecal Microbiota Transplantation on Chronic Functional Constipation and Its Mechanism
Brief Title: Fecal Microbiota Transplantation for Chronic Functional Constipation
Acronym: FMTFCFC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chengdu Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMT-CFC
Record Dates: First submitted 2017-01-03; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Functional Constipation; Intestinal Bacteria Flora Disturbance; Fecal Microbiota Transplantation
Keywords: Chronic Functional Constipation; Intestinal Bacteria Flora Disturbance; Fecal Microbiota Transplantation
MeSH Terms: interventions — Fecal Microbiota Transplantation; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment for part 1 (Active Comparator): Fecal microbiota transplantation and traditional treatments will be used in patients with chronic functional constipation in part 1.
  Interventions: Other: Fecal Microbiota Transplantation
- Placebo for part 2 (Placebo Comparator): The traditional treatments and normal saline will be used in patients with chronic functional constipation in part 2 according to associated guidelines.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Other: Fecal Microbiota Transplantation — Fecal Microbiota Transplantation and the traditional treatments for chronic functional constipation in part 1.
  Other Names: Fecal Microbiota Transplantation(FMT)
  Arms: treatment for part 1
Other: Normal Saline — Normal saline and the traditional treatments for chronic functional constipation in part 2
  Other Names: Normal Saline(NS)
  Arms: Placebo for part 2

SUMMARY:
Chronic functional constipation is a common digestive system disease, the incidence is increasing in recent years.It is reported that the occurrence and development of chronic functional constipation is closely related to imbalance of intestinal flora .Moreover,types and quantity of intestinal flora may be related to intestinal motility. Fecal microbiota transplantation as a new technology to rebuild intestinal flora has been used for several disease，but the clinical efficacy of chronic functional constipation by fecal microbiota transplantation needs to be further explored.

DETAILED DESCRIPTION:
Patients who meet the inclusion crit chronic functional constipation will be separated into two parts depending on acceptation or refuse of Fecal microbiota transplantation.Blood specimen from patients will be collected to analysis intestinal motility.

ELIGIBILITY:
Inclusion criteria:

1. subjects voluntarily participate in the trial and sign informed consent;
2. sex is not limited,ranging from 18 to 75 years old;
3. meet the diagnostic criteria for chronic functional constipation in patients;
4. patients has been ruled out organic diseases of the large intestine within 1 year by colonoscopy or barium enema examination, and stool routine and occult blood examination are normal within 1 month;
5. be able to communicate well with the researchers and follow the verification requirements.

Exclusion criteria:

1. does not meet the diagnostic criteria;
2. with severe primary heart, liver, lung, kidney, blood or affect the survival of serious diseases;
3. severe anemia and severe systemic infection;
4. suspected or indeed have alcohol, drug abuse history;
5. pregnancy or are preparing for pregnancy, and breastfeeding women;
6. Those who are unwilling to accept the research measures or other reasons can not cooperate;
7. due to mental disorders can not give adequate informed consent;
8. Participated in other clinical trials within 3 months before the start of the study;
9. researchers believe that participates are not suitable for other reasons in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events complication rate in all patients in both groups | 3 months

SECONDARY OUTCOMES:
Mean number of bowel movements per week | 4 weeks
Bristol stool scale | 4 weeks
Constipation-related symptoms assessments | 4 weeks
  Constipation-related symptoms were evaluated using the validated Patient Assessment of Constipation Symptoms (PAC-SYM) questionnaire at week 4.
Usage of laxatives or enemas as rescue medication | 4 weeks
Histological changes in the intestinal biopsy in both groups. | 4 weeks
Microbiota composition | 4 weeks
Nitric oxide(NO) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoan Li, Ph.D, Study Chair — First Affiliated Hospital of Chengdu Medical College
Locations (1):
- IEC of Chengdu Medical College, Chendu, China

IPD SHARING:
Plan to Share IPD: No